CLINICAL TRIAL: NCT01191775
Title: A Phase 1 Study of PNT2258 in Patients With Advanced Solid Tumors
Brief Title: A Study of PNT2258 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P06-10091 (PNT2258-01)
Record Dates: First submitted 2010-08-27; First posted 2010-08-31 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2017-01

CONDITIONS: Cancer; Lymphoma; Prostate Cancer; Melanoma
Keywords: Oligonucleotide; DNAi; Oncology; Antineoplastic agent; Lymphoma; PNT2258
MeSH Terms: conditions — Neoplasms; Lymphoma; Prostatic Neoplasms; Melanoma | interventions — PNT100

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PNT2258 (Experimental): PNT2258 is composed of PNT100, a 24-mer oligonucleotide, the active drug substance encapsulated in a liposome.
  Interventions: Drug: PNT2258

INTERVENTIONS:
Drug: PNT2258 — Patients will receive PNT2258 as an intravenous infusion once daily for 5 consecutive days (Days 1-5) of every 21-day cycle (3 weeks). The treatment cycle repeats every 3 weeks for up to 6 cycles in the absence of disease progression, unacceptable toxicity, or patient withdrawal from the study.
  Other Names: PNT-2258

SUMMARY:
This study is sponsored by Sierra Oncology, Inc. formerly ProNAi Therapeutics, Inc. The purpose of this research study is to evaluate the safety of the investigational drug PNT2258 in patients with advance tumors and see how it acts in the body.

DETAILED DESCRIPTION:
This study is an open-label, single-arm, Phase 1 dose-escalation study of PNT2258 in patients with advanced solid tumors for which no standard therapy exists. Patients will receive PNT2258 as an intravenous infusion once daily for 5 consecutive days (Days 1-5) of every 21-day cycle (3 weeks). At first, patients will be treated in single patient cohorts following an accelerated titration design and evaluated for toxicities. After the accelerated portion ends, patients will be treated in cohorts of at least 3 patients at each dose level and evaluated for treatment-related toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, malignant solid tumor (measurable or non-measurable disease) and cannot be a candidate for known regimens or protocol treatments of higher efficacy or priority.
* Recovered to Grade 1 from all acute toxicities of prior therapies, except for residual toxicities, such as alopecia, which do not pose an ongoing medical risk.
* ECOG performance status of 0, 1, or 2.
* At least 18 years of age.
* Patients must have normal organ and marrow function as defined by:

  * Absolute neutrophil count 1,500/µL
  * Platelets 100,000/µL
  * Total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) 2.5 x institutional upper limit of normal (ULN) or 5.0 x ULN in patients with liver metastases
  * Serum creatinine 1.5 x ULN or measured creatinine clearance of 60 mL/min/1.73 m2.
* Negative serum pregnancy test at the time of enrollment for women of child-bearing potential. For men and women of child-producing potential, use of effective contraceptive methods is required during the study.
* Ability to understand the requirements of the study. Must provide written informed consent and authorization of use and disclosure of protected health information. Must agree to abide by the study restrictions and to return for the required assessments.

Exclusion Criteria:

* Received previous anticancer chemotherapy, immunotherapy, radiotherapy or any other investigational therapy in the 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to study entry.
* Receiving any other investigational agents.
* Known brain metastases with the exception of patients with a history of treated brain metastases who are stable for at least 3 months off glucocorticoids and seizure medications.
* Prolongation of QT/QTc interval > 450 milliseconds (ms).
* Known HIV, HBV, or HCV infection.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PNT2258.
* History of allergic reaction to egg or chicken antigens.
* Pregnant or nursing women.
* Uncontrolled intercurrent illness including, but not limited to ongoing or serious active infection, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To determine the safety of PNT2258 in patients with advanced solid tumors | Ongoing
  Safety and tolerability of PNT2258 and the determination of dose-limiting toxicities (DLTs) and the recommended Phase 2 dose

SECONDARY OUTCOMES:
Pharmacokinetic profile of PNT2258 | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Anthony W Tolcher, MD, FRCP(C), Principal Investigator — South Texas Accelerated Research Therapeutics (START)
Locations (1):
- South Texas Accelerated Research Therapeutics (START), San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tolcher AW, Rodrigueza WV, Rasco DW, Patnaik A, Papadopoulos KP, Amaya A, Moore TD, Gaylor SK, Bisgaier CL, Sooch MP, Woolliscroft MJ, Messmann RA. A phase 1 study of the BCL2-targeted deoxyribonucleic acid inhibitor (DNAi) PNT2258 in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2014 Feb;73(2):363-71. doi: 10.1007/s00280-013-2361-0. Epub 2013 Dec 3. PMID 24297683
- See also: Sponsor's Web Site — http://www.sierraoncology.com